CLINICAL TRIAL: NCT04980586
Title: Cheeks Appearance as a Novel Predictor of Obstructive Sleep Apnea The CASA Score Study
Acronym: CASA
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0314
Record Dates: First submitted 2021-07-02; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Obstructive Sleep Apnea; Breathing, Sleep-Disordered; Muscle Weakness; Muscle Disorder; Face; Swallowing Disorder
Keywords: Obstructive sleep apnea; Polysomnography; Orofacial myofunctional disorders; Speech and Language and Hearing Science; Ultrasonography; Muscle Contraction; Muscle Strength; Sleep medicine
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Muscle Weakness; Muscular Diseases; Facies; Deglutition Disorders; Speech; Language | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-OSA Groups: Participants with apnea-hypopnea index < 5 events per hour of sleep.
  Interventions: Diagnostic Test: CASA score protocol to Non-obstructive sleep apnea Group
- Mild OSA Group: Participants with apnea-hypopnea index > 5 < 15 events per hour of sleep.
  Interventions: Diagnostic Test: CASA score protocol to Mild obstructive sleep apnea Group
- Moderate OSA group: Participants with apnea-hypopnea index > 15 < 30 events per hour of sleep.
  Interventions: Diagnostic Test: CASA score protocol to Moderate obstructive sleep apnea Group
- Severe OSA Group: Participants with apnea-hypopnea index > 30 events per hour of sleep.
  Interventions: Diagnostic Test: CASA score protocol to Severe obstructive sleep apnea Group

INTERVENTIONS:
Diagnostic Test: CASA score protocol to Non-obstructive sleep apnea Group — CASA score observe the cheeks appearance: volume of the cheeks (0, 1, 2 or 3) and flaccidity, (0, 1, 2 or 3). The final score is volume + flaccidity score to have the CASA score (0-6). A photography was captured to enable the blinded evaluation of three evaluators of each participant. Ultrasonography was positioned in the face of the participant and slide to capture the muscle image (masseter muscle, buccinator and the tongue). Tongue and cheeks pressure were assessed with a device with a small bulb. Inside the mouth in the tongue, the participant is instructed to press the bulb against the hard palate. In the cheeks, the bulb is placed between the cheek and the teeth and the participant press the bulb with the cheek. Swallowing evaluation with an endoscope that enters in the nose of the participant to observe the the oropharynx; while the participant is eating liquid consistency, pureed consistency and solid food.
  Other Names: Photography registers; Ultrasonography in Specific Orofacial Muscles by BodyMetrix device; Tongue and Cheeks Pressure Evaluation by Iowa Oral Performance Instrument Medical Device; Swallowing evaluation by Endoscopy
  Groups: Non-OSA Groups
Diagnostic Test: CASA score protocol to Mild obstructive sleep apnea Group — CASA score observe the cheeks appearance: volume of the cheeks (0, 1, 2 or 3) and flaccidity, (0, 1, 2 or 3). The final score is volume + flaccidity score to have the CASA score (0-6). A photography was captured to enable the blinded evaluation of three evaluators of each participant. Ultrasonography was positioned in the face of the participant and slide to capture the muscle image (masseter muscle, buccinator and the tongue). Tongue and cheeks pressure were assessed with a device with a small bulb. Inside the mouth in the tongue, the participant is instructed to press the bulb against the hard palate. In the cheeks, the bulb is placed between the cheek and the teeth and the participant press the bulb with the cheek. Swallowing evaluation with an endoscope that enters in the nose of the participant to observe the the oropharynx; while the participant is eating liquid consistency, pureed consistency and solid food.
  Other Names: Photography registers; Ultrasonography in Specific Orofacial Muscles by BodyMetrix device; Tongue and Cheeks Pressure Evaluation by Iowa Oral Performance Instrument Medical Device; Swallowing evaluation by Endoscopy
  Groups: Mild OSA Group
Diagnostic Test: CASA score protocol to Moderate obstructive sleep apnea Group — CASA score observe the cheeks appearance: volume of the cheeks (0, 1, 2 or 3) and flaccidity, (0, 1, 2 or 3). The final score is volume + flaccidity score to have the CASA score (0-6). A photography was captured to enable the blinded evaluation of three evaluators of each participant. Ultrasonography was positioned in the face of the participant and slide to capture the muscle image (masseter muscle, buccinator and the tongue). Tongue and cheeks pressure were assessed with a device with a small bulb. Inside the mouth in the tongue, the participant is instructed to press the bulb against the hard palate. In the cheeks, the bulb is placed between the cheek and the teeth and the participant press the bulb with the cheek. Swallowing evaluation with an endoscope that enters in the nose of the participant to observe the the oropharynx; while the participant is eating liquid consistency, pureed consistency and solid food.
  Other Names: Photography registers; Ultrasonography in Specific Orofacial Muscles by BodyMetrix device; Tongue and Cheeks Pressure Evaluation by Iowa Oral Performance Instrument Medical Device; Swallowing evaluation by Endoscopy
  Groups: Moderate OSA group
Diagnostic Test: CASA score protocol to Severe obstructive sleep apnea Group — CASA score observe the cheeks appearance: volume of the cheeks (0, 1, 2 or 3) and flaccidity, (0, 1, 2 or 3). The final score is volume + flaccidity score to have the CASA score (0-6). A photography was captured to enable the blinded evaluation of three evaluators of each participant. Ultrasonography was positioned in the face of the participant and slide to capture the muscle image (masseter muscle, buccinator and the tongue). Tongue and cheeks pressure were assessed with a device with a small bulb. Inside the mouth in the tongue, the participant is instructed to press the bulb against the hard palate. In the cheeks, the bulb is placed between the cheek and the teeth and the participant press the bulb with the cheek. Swallowing evaluation with an endoscope that enters in the nose of the participant to observe the the oropharynx; while the participant is eating liquid consistency, pureed consistency and solid food.
  Other Names: Photography registers; Ultrasonography in Specific Orofacial Muscles by BodyMetrix device; Tongue and Cheeks Pressure Evaluation by Iowa Oral Performance Instrument Medical Device; Swallowing evaluation by Endoscopy
  Groups: Severe OSA Group

SUMMARY:
Cheeks appearance is a screening tool developed based on cheeks observation to identify volume, flaccidity or both to predict people with probable obstructive sleep apnea.

DETAILED DESCRIPTION:
Cheeks Appearance for Sleep Apnea (CASA score) is a screening tool developed to observe adults people cheeks appearance to identify volume, being 0 for no volume, 1 for mild volume, 2 for moderate volume and 3 for severe volume; or flaccidity, being 0 for no flaccidity, 1 for mild flaccidity, 2 for moderate flaccidity and 3 for severe flaccidity. In the end of CASA score screening we sum up the score of volume with the score and the flaccidity score to reach the CASA score, the final result that can range from 0 to 6 points.

This study was applied in three moments, being the first one only the application of CASA score and a facial imaging to facilitate the replicability. The data collection and enrollment of 248 participants were made in a sleep private clinic in participants undergoing polysomnography. All this part of data collection was applied for a 3 months period. This first part was the validation of CASA score protocol with internal validity.

The second part was carried out 1 year after in which all participants enrolled were evaluated by CASA score and facial imaging, as the first part, in a sleep private clinic while doing polysomnography. Additionally, procedures such as ultrasonography images of specific orofacial muscles, followed by tongue and cheeks pressure evaluation were carried out just after the CASA score and facial imaging based on photography registers. In this second part, others 71 participants were recruited.

The third and last part was a case-control study in which 20 of the 71 anterior part of the data collection were invited to take part in the last part of the study, that was the fiberoptic endoscopic evaluation of swallowing, so 10 non obstructive sleep apnea participants and 10 obstructive sleep apnea participants were chosen and invited, 19 accepted and carried out the last part. This last part was underwent in an outpatient clinic of an otorhinolaryngologist or ear, nose and throat physician (ENT) with a Speech and Language Therapist (SLT).

Description of the methods:

Ultrasonography was made with a portable device which was positioned in the face of the participant and slide for the direction needed to capture the image of the muscle targeted like masseter, buccinator and tongue. Those were the three muscles evaluated by the ultrasonography exam.

Tongue and cheeks pressure evaluation was made with IOPI medical equipment which had a small bulb coupled in the device and its bulb was positioned inside the mouth of the participant in the tongue and the participant was instructed to press as hard as he could against the hard palate. In the cheeks was positioned in the oral vestibule between the cheek and the teeth, and the pressure was applied by the cheeks.

Fiberoptic endoscopic evaluation of swallowing (FEES): a micro camera of a endoscopy was inserted in the participant nose to look the nasopharynx and oropharynx. The fiberoptic was kept in the nasopharynx to see the participant eating, first a liquid consistency (5 and 10 ML), pureed consistency (5 and 10 ML) and solid food (half cracker and 1 whole cracker). The whole exam lasted 15 to 20 minutes, maximum.

ELIGIBILITY:
Inclusion Criteria:

* Sleep complaints
* 18 years old or older
* Undergoing polysomnography in the private sleep clinic

Exclusion Criteria:

* Previous OSA diagnose
* Severe comorbidities such as neurologic diseases or others condition that could cause facial edema or facial deformities
* Facial hair that could difficult the facial landmarks visualization
* Previous facial surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over 18 years old with sleep complaints undergoing he polysomnography in the private sleep clinic during the data collection period.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Cheeks appearance | Immediately after the evaluation
  Identify cheeks volume and cheeks flaccidity, choose the correspondent number of volume and flaccidity 0, 1, 2 or 3, sum up both and reach the final score that is CAS score.

SECONDARY OUTCOMES:
Thickness evaluation of specific orofacial muscles | Immediately after the evaluation
  Identify the thickness of the masseter, the buccinator and the tongue of each participant and compare with cheeks appearance outcome
Tongue and Cheeks pressure | Immediately after the evaluation
  Identify the maximum pressure of the tongue and the maximum pressure of the cheek (both sides) and compare with cheeks appearance and thickness evaluation outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Denis Martinez, Study Chair — Hospital de Clinicas de Porto Alegre (HCPA)
Locations (1):
- Hospital de Clínicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agha B, Johal A. Facial phenotype in obstructive sleep apnea-hypopnea syndrome: a systematic review and meta-analysis. J Sleep Res. 2017 Apr;26(2):122-131. doi: 10.1111/jsr.12485. Epub 2016 Dec 26. PMID 28019049
- [Background] Harrington JJ, Avidan AY. Treatment of sleep disorders in elderly patients. Curr Treat Options Neurol. 2005 Sep;7(5):339-52. doi: 10.1007/s11940-005-0027-x. PMID 16079039
- [Background] Guimaraes KC, Drager LF, Genta PR, Marcondes BF, Lorenzi-Filho G. Effects of oropharyngeal exercises on patients with moderate obstructive sleep apnea syndrome. Am J Respir Crit Care Med. 2009 May 15;179(10):962-6. doi: 10.1164/rccm.200806-981OC. Epub 2009 Feb 20. PMID 19234106
- [Background] Lee RW, Chan AS, Grunstein RR, Cistulli PA. Craniofacial phenotyping in obstructive sleep apnea--a novel quantitative photographic approach. Sleep. 2009 Jan;32(1):37-45. PMID 19189777
- [Background] Perri RA, Kairaitis K, Cistulli P, Wheatley JR, Amis TC. Surface cephalometric and anthropometric variables in OSA patients: statistical models for the OSA phenotype. Sleep Breath. 2014 Mar;18(1):39-52. doi: 10.1007/s11325-013-0845-0. Epub 2013 Apr 13. PMID 23584845
- [Background] Lee RW, Petocz P, Prvan T, Chan AS, Grunstein RR, Cistulli PA. Prediction of obstructive sleep apnea with craniofacial photographic analysis. Sleep. 2009 Jan;32(1):46-52. PMID 19189778
- [Background] Kim AM, Keenan BT, Jackson N, Chan EL, Staley B, Poptani H, Torigian DA, Pack AI, Schwab RJ. Tongue fat and its relationship to obstructive sleep apnea. Sleep. 2014 Oct 1;37(10):1639-48. doi: 10.5665/sleep.4072. PMID 25197815
- [Background] Yoshikawa M, Yoshida M, Tsuga K, Akagawa Y, Groher ME. Comparison of three types of tongue pressure measurement devices. Dysphagia. 2011 Sep;26(3):232-7. doi: 10.1007/s00455-010-9291-3. Epub 2010 Jul 11. PMID 20623302
- [Background] Valbuza JS, de Oliveira MM, Zancanella E, Conti CF, Prado LB, Carvalho LB, do Prado GF. Swallowing dysfunction related to obstructive sleep apnea: a nasal fibroscopy pilot study. Sleep Breath. 2011 May;15(2):209-13. doi: 10.1007/s11325-010-0474-9. Epub 2011 Jan 13. PMID 21229321
- [Background] Prikladnicki A, Martinez D, Brunetto MG, Fiori CZ, Lenz MDCS, Gomes E. Diagnostic performance of cheeks appearance in sleep apnea. Cranio. 2018 Jul;36(4):214-221. doi: 10.1080/08869634.2017.1376426. Epub 2017 Sep 21. PMID 28933667
- [Background] Smith-Ryan AE, Fultz SN, Melvin MN, Wingfield HL, Woessner MN. Reproducibility and validity of A-mode ultrasound for body composition measurement and classification in overweight and obese men and women. PLoS One. 2014 Mar 11;9(3):e91750. doi: 10.1371/journal.pone.0091750. eCollection 2014. PMID 24618841
- [Derived] Prikladnicki A, Gomes E, Cortes Reis Sousa LC, Goncalves SC, Martinez D. Cheeks appearance as a novel predictor of obstructive sleep apnea: the CASA score study. J Clin Sleep Med. 2024 Jun 1;20(6):879-885. doi: 10.5664/jcsm.11022. PMID 38217481
- See also: Our first study in diagnostic accuracy in obstructive sleep apnea and the basis to this study. — https://pubmed.ncbi.nlm.nih.gov/28933667/